CLINICAL TRIAL: NCT02135068
Title: Preventing Hypoglycemia During Exercise With Proactive Snacking on Closed Loop
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jennifer Sherr, Instructor, Yale University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1403013588; T32DK063703 (NIH)
Record Dates: First submitted 2014-04-16; First posted 2014-05-09 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; closed loop insulin delivery systems; exercise; hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoglycemia | interventions — Drug Delivery Systems; Snacks; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CL and exercise with proactive snacking (Experimental): Subject will consume oral glucose prior to starting exercise regimen while on the Medtronic MiniMed Closed Loop (CL) System
  Interventions: Device: Medtronic MiniMed Closed Loop (CL) System; Other: Snacking
- CL and exercise without proactive snacking (Active Comparator): Subject will not consume oral glucose prior to starting exercise regimen while on the Medtronic MiniMed Closed Loop (CL) System
  Interventions: Device: Medtronic MiniMed Closed Loop (CL) System

INTERVENTIONS:
Device: Medtronic MiniMed Closed Loop (CL) System — The Medtronic MiniMed Closed Loop (CL) System is an investigational system that uses some commercially available products. An investigational Enlite 2 glucose sensor measures the sensor glucose. The glucose sensor signal is sent to the insulin pump. From the insulin pump the sensor glucose is sent through the translator, which then relays the signal on to a controller. An Android Mobile Device (off the shelf) has the control algorithm installed. This device is known as the controller. The controller serves as the control center for the Android system, receiving data from the sensor and pump components, feeding the data to its control algorithm, issuing delivery commands to the pump to apply the algorithm's recommend therapy, and providing a means to monitor the system.
Other: Snacking — Up to 45 g of oral glucose via Gatorade
  Other Names: Oral glucose
  Arms: CL and exercise with proactive snacking

SUMMARY:
This study is designed to look at how snacking during exercise may help prevent low blood sugars while subjects are on the "closed loop artificial pancreas." This system uses a continuous glucose sensor, an insulin pump, and a computer program that automatically determines how much insulin to give based on the sensor glucose level.

DETAILED DESCRIPTION:
This study will be a randomized cross-over study as subjects will be studied under both study conditions - Closed Loop (CL) alone vs. CL + proactive snacking protocol). Differences in the nadir blood glucose levels during exercise between the two study conditions will be the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 13-45 years
2. Clinical diagnosis of T1D (formal antibody and/or genetic testing will not be required)
3. Duration of T1D ≥ 1 year
4. HbA1c ≤ 9 %
5. Treated with continuous subcutaneous insulin infusion (pump) for at least 3 months
6. Body weight > 40 kg (to accommodate phlebotomy)
7. Able to tolerate a 75-minute exercise period of moderate intensity
8. Be willing to wear 2 subcutaneous glucose sensors (placed under the skin like a pump site) simultaneously during the inpatient portions of this study.
9. Be in good general health without other acute or chronic illness that in the judgment of the investigator could interfere with the study or jeopardize subject safety
10. Normal hematocrit
11. Able to give consent (for children <18 years, permission from parents and subject assent will be required)
12. Female subjects of reproductive potential must be abstinent or consistently using appropriate family planning methods.

Exclusion Criteria:

1. Insulin resistant (defined as requiring > 1.5 units/kg/day at time of study enrollment)
2. Presence of any medical or psychiatric disorder that may interfere with subject safety or study conduct
3. Use of any medications (besides insulin) known to effect blood glucose levels, including oral or other systemic glucocorticoid therapy. Inhaled, intranasal, or rectal corticosteroid use is allowed along as not given within 2 weeks of the closed loop admissions. Use of topical glucocorticoids is allowable as long as affected skin area does not overlap with study device sites.
4. Subjects using herbal supplements will be excluded, due to the unknown effects of these supplements on glucose control
5. History of hypoglycemic seizure within last 3 months
6. Female subjects who are pregnant, lactating, or unwilling to be tested for pregnancy

Ages: 13 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Nadir blood glucose levels during exercise | 75 minutes
  Difference in the nadir blood glucose levels during exercise between the two study conditions: Closed Loop alone vs. Closed Loop+ snacking.

SECONDARY OUTCOMES:
Episodes of hypoglycemia (blood glucose <60mg/dL) during exercise | 75 minutes
  Percentage of subjects that required treatment for hypoglycemia during the exercise period between the two study conditions
Mean reduction in blood glucose during exercise | 75 minutes
  Mean Reduction in blood glucose from baseline blood glucose during exercise
Mean time blood glucose in target during exercise | 75 minutes
  Comparison of the mean time blood glucose levels were between 70-180mg/dL during exercise between the two study conditions
Mean time blood glucose levels are in target during the overnight period | 17 hours
  Comparison of the mean time blood glucose levels are in target (70-180mg/dL) during the overnight period after mid-afternoon exercise.
Mean glucose values | 12 hours
  Comparison of the mean daytime and nighttime glucose values
Mean 24- hour glucose levels | 24 hours
  Comparison of the mean 24- hour glucose levels
insulin delivery during CL therapy | 24 hours
  Differences between insulin delivery during CL therapy during the two study conditions (pro-active snacking vs. no snacking) will be assessed.
Incremental meal-related glucose Area Under the Curve | 24 hours
  Assessment of incremental meal related glucose area under the curve will be conducted.
Nadir glucose levels following the meals | 24 hours
  Nadir glucose levels following meals will be compared between the two study conditions
Area under the curve meal-related plasma insulin level excursion following meals | 24 hours
  Area under the curve meal-related insulin excursion following meals.
Nadir glucose levels overnight | 12 hours
  Difference between nadir glucose levels between the two study conditions will be assessed.
Mean absolute relative difference (MARD) for each sensor | 24 hours
  Calculation and comparison of the mean absolute relative difference for each sensor will be performed and comparisons between accuracy of the sensors will be done.
Mean daytime and nighttime glucose values | 24 hours
  Comparison of the mean daytime and nighttime glucose levels

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Sherr, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States